CLINICAL TRIAL: NCT05007236
Title: A Randomized, Double-blind, Placebo-controlled, Phase 2 Study to Evaluate the Efficacy and Safety of Oral RP7214, a DHODH Inhibitor, in Patients With Symptomatic Mild SARS-CoV-2 Infection.
Brief Title: Study to Evaluate the Efficacy and Safety of Oral RP7214, a DHODH Inhibitor, in Patients With Symptomatic Mild COVID-19 Infection.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rhizen Pharmaceuticals SA (Industry)
Collaborators: Incozen Therapeutics Pvt Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RP7214-2101
Record Dates: First submitted 2021-08-09; First posted 2021-08-16 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2022-04

CONDITIONS: SARS-CoV-2 Infection
MeSH Terms: conditions — COVID-19 | interventions — RP7214; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RP7214 + Standard of care (SOC) (Experimental)
  Interventions: Drug: RP7214 + Standard of care (SOC)
- Placebo + Standard of care (SOC) (Placebo Comparator)
  Interventions: Drug: Placebo + Standard of care (SOC)

INTERVENTIONS:
Drug: RP7214 + Standard of care (SOC) — RP7214 tablets will be administered orally twice a day for 14 days
  Arms: RP7214 + Standard of care (SOC)
Drug: Placebo + Standard of care (SOC) — Placebo will be administered orally twice a for 14 days
  Arms: Placebo + Standard of care (SOC)

SUMMARY:
This is a randomized, double-blind, placebo-controlled study of RP7214 in patients with symptomatic mild SARS-CoV-2 infection, having at least one high-risk feature (e.g., age > 60 years, hypertension, diabetes mellitus, chronic lung disease, chronic kidney disease, liver disease, cerebrovascular disease, obesity, cancer) for developing severe Covid-19 illness.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide informed consent.
2. Males and females of ≥ 18 years of age
3. Patient with mild COVID-19 infection having ≥ 1 symptoms.
4. Laboratory confirmed Covid-19 infection by Reverse Transcription Polymerase Chain Reaction (RT-PCR) in nasopharyngeal sample (within 72 hours prior to randomization).
5. Patient should have at least one pre-existing high-risk feature for developing severe Covid-19 illness.
6. Ability to swallow and retain oral medication.
7. Male patient who is surgically sterile, or who is willing to agree to use a contraceptive measure.
8. Women of childbearing potential should be willing to use a medically acceptable method of contraception.
9. Willing to receive telephone calls or have videoconferences with study team personnel.
10. Willing and able to understand the nature of this study, comply with the study procedures and follow-up procedures as per the study protocol.

Exclusion Criteria:

1. Patient with asymptomatic Covid-19 infection.
2. Patient who has experienced the onset of any of Covid-19 symptoms > 5 days at the time of randomization.
3. Moderate to Severe COVID-19 infection
4. Patient with Covid-19 re-infection
5. Subjects who are severely immunocompromised
6. Subjects with autoimmune diseases
7. Patients with any bleeding disorder e.g., hemophilia and von Willebrand disease.
8. Current use of other DHODH inhibitors including teriflunomide or leflunomide.
9. Patients who are on or immediately require Covid-19 directed treatment such as antivirals, immunomodulatory treatment, convalescent plasma, oral/ intravenous steroids, or monoclonal antibodies at the time of screening.
10. Patients who have had received one or two doses of vaccine for Covid-19.
11. Patients participating in another clinical study or use of any investigational product within 4 weeks or 5 half-lives of the drug, whichever is longer, before the date of dosing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2021-09-20 (Actual); Primary Completion 2022-03-25 (Actual); Study Completion 2022-03-25 (Actual)

PRIMARY OUTCOMES:
Proportion of patients requiring Covid-19 related hospitalization by Day 15. | 15 days

SECONDARY OUTCOMES:
Change from baseline in SARS-CoV-2 viral load at Days 3, 7 and 15 by quantitative RT-PCR test | 15 days
Time to symptom resolution in patients receiving RP7214 as compared to placebo | 15 days
Proportion of patients demonstrating symptom resolution | 15 days
Time to symptom improvement in patients receiving RP7214 as compared to placebo | 15 days
Proportion of patients demonstrating symptom improvement | 15 days
Adverse Events (AEs) as assessed by laboratory tests, vital signs and physical examination. | 15 days
Change in the disease-specific inflammatory markers (Ferritin, C-reactive protein (CRP), D-dimer, neutrophil to lymphocyte/CD8+ ratio, LDH, IL-6) as compared to baseline. | 15 days

CONTACTS AND LOCATIONS:
Locations (16):
- India (16):
  - Citizen Hospital, Bangalore
  - Madhu Superspeciality Hospital & Research Center, Bangalore
  - Rajalakshmi Hospital & Research Center, Bangalore
  - Panimalar medical college hospital and research institute, Chennai
  - Maharaja Agrasen Superspeciality Hospital, Jaipur
  - Nil Ratan Sircar Medical College and Hospital, Kolkata
  - Malabar Medical College, Kozhikode
  - BAJ RR Hospital & Research center, Mumbai
  - DEC Healthcare Hospital, Nellore
  - Vijaya Super specialty Hospital, Nellore
  - Jivanrekha Multispeciality Hospital, Pune
  - PCMC'S PGI Yashwantrao Chavan Memorial Hospital, Pune
  - Sant Dnyaneshwar Hospital (Accord Multispeciality Hospital), Pune
  - Govt General Hospital, Srikakulam
  - Great Eastern medical school and hospital, Srikakulam
  - King George Hospital, Visakhapatnam

IPD SHARING:
Plan to Share IPD: No